CLINICAL TRIAL: NCT06177249
Title: Evaluation With Rabies Vaccine (Vero Cell) of Two Different Immune Procedure in the Healthy Crowd the Immunogenicity and Safety of Randomized, Blinded, Similar Vaccine Against Ⅲ Phase of Clinical Trials
Brief Title: To Evaluate the Immunogenicity and Safety of Two Different Immunization Schedules of Rabies Vaccine (Vero Cell)
Acronym: rabies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hualan Biological Bacterin Co. Ltd. (Industry)
Collaborators: Henan Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2014L00266
Record Dates: First submitted 2023-12-07; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2015-03

CONDITIONS: Rabies Human
Keywords: Antibody Titer

STUDY DESIGN:
Intervention Model Description: Lyophilized rabies vaccine for human use (Vero cell) and control vaccine
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental vaccines and vaccine (Active Comparator): A total of 1956 subjects were randomly divided into three groups at a ratio of 1:1:1, 652 subjects in each group were vaccinated with the test vaccine or the control vaccine on a schedule of 0, 3, 7, 14, 28 days (a total of 5 doses). Blood samples were collected from the subjects for antibody detection on 0, 7/14, 35/42 days, respectively.
  Interventions: Biological: Control vaccine; Biological: Experimental vaccine
- experimental vaccines (Active Comparator): An additional group of 652 people received the trial vaccine in a 0 -, 7 -, and 21-day schedule (two first doses for a total of four doses). Blood samples were collected at 0, 7/14 and 35/42 days for antibody detection, and all subjects were systematically observed for safety.
  Interventions: Biological: Experimental vaccine

INTERVENTIONS:
Biological: Control vaccine — A group of 652 subjects were vaccinated with the control vaccine at 0, 3, 7, 14 and 28 days (5 doses in total). Blood samples were collected from the subjects at 0, 7/14 and 35/42 days for antibody detection.
  Arms: Experimental vaccines and vaccine
Biological: Experimental vaccine — A total of 652 subjects received 5 doses of the vaccine at 0, 3, 7, 14 and 28 days. Blood samples were collected on 0, 7/14 and 35/42 days for antibody detection.

SUMMARY:
To evaluate the safety and immunogenicity of lyophilized human rabies vaccine (Vero cell) developed by Hualan Biological in healthy people aged 9 to 65 years with two different immunization schedules.

DETAILED DESCRIPTION:
The trial to assess the rabies vaccine (Vero cells) in healthy group of 9 ~ 65 years old after inoculation, the first dose after 14 days and 14 days after inoculation 5 agent group turn antibody positive rate of bad effect on 5 agent in the control group; The safety profile, seroconversion rate, and geometric mean concentration of the four-dose vaccine were noninferior to those of the five-dose regimen at 14 days after the first dose. More people aged 9-65 in the first agent free after 7 days, 14 days and 14 days after inoculation, 5 patients and 5 doses in the control group, four patients and 5 doses group antibody positive rate, GMC and GMC growth multiples have differences. To evaluate whether the seroconversion rate of subjects in the 4-dose experimental group reached 100% 14 days after the whole course of vaccination.

ELIGIBILITY:
Inclusion Criteria:

* 9 to 65 years old healthy residents;
* volunteered for the experiment and signed informed consent;
* the subjects or their guardians can comply with the requirements of the clinical trial protocol;
* have not received rabies vaccination at any time;
* nearly six months has not been mammals bite, scratch;
* not participating in clinical trials of other drugs;
* No use of human immunoglobulin or other products in the past six months.

Exclusion Criteria:

First needle exclusion:

* have allergies, convulsions, seizures, mental and nervous system, such as history, or family history of epilepsy;
* Allergic to the main ingredient of the investigational vaccine;
* known to people with poor immune function damage or the tumor, spleen;
* Axillary temperature >38.0℃ within 7 days due to acute febrile illness;
* Patients with axillary body temperature > 37.0℃;
* Severe chronic diseases such as congenital malformation, developmental disorder or severe cardiovascular disease, diabetes mellitus, hypertension that cannot be stabilized by drugs, liver and kidney diseases, and malignant tumors;
* patients with acute and chronic infectious diseases, active infections, severe asthma, infectious skin diseases;
* pregnant and lactating women; Any circumstances that the investigator believes may affect the assessment of the trial.

Subsequent needle exclusions:

* any serious adverse event causally related to vaccination;
* new findings that meet the "first dose exclusion criteria";
* the researchers think that may affect test evaluation of any situation.

Ages: 9 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1956 (Actual)
Dates: Start 2015-03-15 (Actual); Primary Completion 2015-12-16 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
1956 subjects accept the observation of local adverse reaction according to Guidelines for grading standard of adverse reaction of clinical trial of vaccine used for prevention | Every needle 30 days after vaccination
  Tenderness, pruritus, induration, redness, swelling and its degree of size and disturbance of body activity at the inoculation site
1956 subjects accept the observation of local adverse reaction according to Guidelines for grading standard of adverse reaction of clinical trial of vaccine used for prevention | Vaccinations 31 days to 180 days
  Tenderness, pruritus, induration, redness, swelling and its degree of size and disturbance of body activity at the inoculation site
1956 subjects accept the observation of systemic adverse reactions according to Guidelines for grading standard of adverse reaction of clinical trial of vaccine used for prevention. | Every needle 30 days after vaccination
  Fever, allergy, headache, fatigue, nausea and vomiting, diarrhea, muscle pain, arthralgia and so on were observed
1956 subjects accept the observation of systemic adverse reactions according to Guidelines for grading standard of adverse reaction of clinical trial of vaccine used for prevention. | Vaccinations 31 days to 180 days
  Fever, allergy, headache, fatigue, nausea and vomiting, diarrhea, muscle pain, arthralgia and so on were observed

SECONDARY OUTCOMES:
The immunogenicity was tested by immunofluorescence staining | 5 agent group gathering subjects were 0, 7, 14, 42 days of blood samples
  The rabies virus antibody was detected by immunofluorescence focus method. The positive rate was defined as the serum antibody concentration ≥0.5IU/ml
The immunogenicity was tested by immunofluorescence staining | Blood samples were collected on day 0, 7, 14 and 35 in the 4-dose group
  The rabies virus antibody was detected by immunofluorescence focus method. The positive rate was defined as the serum antibody concentration ≥0.5IU/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Xia Shengli, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No